CLINICAL TRIAL: NCT05961644
Title: Safety and Efficacy of Subcutaneous Cladribine for Nonrelapsing, Secondary Progressive Multiple Sclerosis (CLASP-MS): a Randomized, Placebo-controlled, Double-blind, Phase 2 Study.
Brief Title: Cladribine vs Placebo for Non-active Progressive Multiple Sclerosis (CLASP-MS).
Acronym: CLASP-MS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Psychiatry and Neurology, Warsaw (Other)
Collaborators: Nalecz Institute of Biocybernetics and Biomedical Engineering, Polish Academy of Sciences (Other); Mossakowski Medical Research Centre Polish Academy of Sciences (Other); Poznan University of Medical Sciences (Other); Military Institute of Aviation Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 504-15-021-21003; 2022-000036-32 (EudraCT Number); 2021/ABM/02/00002/P/02 (Other Grant/Funding Number: Medical Research Agency in Poland); DBL.474.362.2022 (Registry Identifier: Office for Registration of Medicinal Products)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis
Keywords: Cladribine; Multiple Sclerosis Secondary Progressive; Brain Volume; Quantitative Susceptibility Mapping; Magnetic Resonance Imaging; Cognitive assessment
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Drug: Cladribine at a dose of 1.8 mg/kg of body weight. Cladribine will be given subcutaneously over 6 visits every 5-6 weeks.
  Interventions: Drug: Cladribine Subcutaneous Injection
- Control (Placebo Comparator): Comparator: Placebo matched to the subcutaneous injection of cladribine.
  Interventions: Drug: 0.9% Chloride Injection Sodium

INTERVENTIONS:
Drug: Cladribine Subcutaneous Injection — Cladribine subcutaneous injection, 10 mg daily, for 2-3 consecutive days (depending on individual dose)
  Other Names: Cladribine Solution
  Arms: Experimental
Drug: 0.9% Chloride Injection Sodium — 0.9% sodium chloride injected subcutaneously, 10 ml daily, for 2-3 consecutive days
  Arms: Control

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of subcutaneously administered cladribine versus placebo to stop inflammation and treat disease progression of non-active secondary progressive multiple sclerosis.

Multiple sclerosis is an inflammatory disease of the central nervous system. In most patients, it starts with a relapsing course (RMS) which is caused by acute inflammatory lesions in the brain and spinal cord. RMS transforms at later stages into progressive disease (secondary progressive MS). Currently approved disease-modifying treatments are effective in reducing clinical relapses and brain and spinal lesions visible in MR, but they perform poorly in preventing disease progression and overall disability accumulation. The growing evidence shows that disease progression partially depends on chronic inflammation present in the CNS. Drugs, which may cross the blood-brain barrier and reach inflammatory cells residing in the CNS might be effective in this stage of the disease. Cladribine is one of the DMT approved for RMS. It is a synthetic purine analog with selective lymphocyte toxicity, which enter the CNS and is found in cerebrospinal fluid. In patients treated with cladribine, the oligoclonal bands tend to disappear proving that neuroinflammation is diminished.

The participants of this clinical trial with the later non-active stage of MS are enrolled to be treated with cladribine subcutaneously or a non-active comparator (placebo) for 6 months and followed for the next 2 years, with an MRI scan and clinical evaluation every 6 months. The main questions it aims to answer are if in the non-active stage of MS cladribine is potent to lessen brain volume loss and if it is potent to attenuate inflammation in the CNS.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multi-center, phase 2 study of subcutaneous cladribine in non-relapsing, secondary progressive multiple sclerosis. Eligible patients will be randomly allocated in a 1:1 ratio to receive either placebo or subcutaneous cladribine at a dose of 1.8 mg/kg of body weight. The study will consist of three periods: screening, treatment, and follow-up. During the screening, the investigators will assess patient eligibility. During the treatment, cladribine will be given over 6 visit every 5-6 weeks. During the follow-up of 96 weeks, safety and efficacy assessments will be carried out on five visits: the first visit will take place 4 weeks after the last cladribine dose, and the remaining visits will take place every 24 weeks.

There will a rescue option of unblinding and treatment with a full dose of cladribine (cladribine arm) or approved medications (placebo arm) for patients with a severe relapse or ≥ 2 non-severe relapses after enrolment or with a substantial neuroimaging disease activity ≥ 4 Gd+ lesions in any scan, ≥ 3 Gd+ lesions in any two scans, ≥ 2 Gd+ lesions in any three scans, or ≥ 9 new/enlarging T2 lesions on any scan compared with baseline).

All raters will be blinded to treatment allocation. All neuroimaging examinations will be evaluated at a central neuroimaging unit by investigators blinded to treatment allocation.

Study type: interventional (clinical trial) Planned enrolment: 188 patients Allocation: randomized Masking: Double (Participant, Investigator) Primary purpose: Treatment Start Date: October 2022

Study design: The study aims to assess the safety and efficacy of subcutaneous cladribine in patients with SPMS who have not experienced relapses over a year and with or without active lesions on neuroimaging. The study will be randomized, placebo-controlled, and double blind. Because no treatment is approved for inactive SPMS, placebo was chosen as the comparator. Patients receiving other treatments for SPMS or immunosuppressant will not be included.

The study will consist of the following phases:

1. Screening phase (about 4 weeks)
2. Treatment phase, patients will be randomized 1:1 ratio of either cladribine 1,8mg/kg or placebo (30 weeks)
3. Follow-up phase , patients will be followed every 24 weeks for up to 122 weeks for safety and efficacy of the treatment;

Patients: The group of 188 patients fulfilling inclusion criteria and not-fulfilling exclusion criteria will enrolled to the study. All patient has to sign written informed consent form approved by Ethics Committee.

Blinding: Randomization and blinding will be done by "dual assessor" approach . Every site will have two teams of blinded and blinded investigators . The blinded investigators include Principal or treating investigators and rating investigators, as well as blinded treating nurse. The unblinded team includes: Randomizing investigator responsible also for laboratory assessment and unblinded nurse/pharmacist responsible for preparing drugs.

Intervention:

Experimental arm Drug: Cladribine at a dose of 1.8 mg/kg of body weight. Cladribine will be given subcutaneously over 6 visits every 5-6 weeks.

Comparator: Placebo matched to the subcutaneous injection of cladribine.

Follow-up: Patients will be assessed and baseline visit, and every 24 weeks over 24 months since the last dose of the interventional drug. The evaluations include:

1. Medical history, concomitant medication, relapse history
2. Physical examination, neurological examination
3. Clinical assessment: EDSS, T25FWT, 9-HPT,
4. MsQoL and CSSR scale
5. MRI of head and spinal cord (baseline, every 6 months for head and every 12 months for spinal cord)
6. Laboratory and biomarkers evaluation (hematology, coagulation, HIV serology, Hepatitis virus B and C serology, tuberculosis tests (Quantiferron test if necessary), ,

The primary end point will be percentage brain volume change between the last dose (week 24) and end of study (week 122). The primary endpoint was selected based on the widely discussed indications for designing studies in the SPMS. The main secondary clinical end points will assess the change in neurological function on the Expanded Disability Status Scale, Timed 25 Foot Walk, and 9-Hole Peg Test, which measures upper limb function. The change in cognitive function will be assessed with various neuropsychological tests. The main secondary neuroimaging end points will include change in the number of contrast-enhancing lesions, the number of T1-hypointesne lesions ("black holes"), and the volume of T2 lesions. The main exploratory end point will be the change in QSM rim+ lesions on brain neuroimaging; these lesions are markers of chronic, smoldering neuroinflammation that may take place behind an intact blood-brain barrier. Change in the concentrations of neurofilament light chain and glial fibrillary acidic protein, which are markers of brain tissue damage, will be main laboratory end points. An exploratory analysis of inflammatory protein biomarkers will be carried out in serum and cerebrospinal fluid of a selected patients (Luminex). The study will assess the safety of cladribine and its effect on quality of life.

The proposed intervention is well supported by the current evidence. Cladribine is among the few drugs that penetrate an intact blood-brain barrier, which allows action on lymphocytes resident in the central nervous system. The study will assess whether cladribine slows down disease progression clinically and it will use the best currently available indicators of disease progression: brain and cervical cord atrophy and the number of demyelinating lesions. Additionally, it will be assessed whether the presence of QSM rim+ lesions is associated with disease course and the therapeutic effect of cladribine. For example, a reduction in the number of these lesions during cladribine treatment would supports an action of the drug behind the blood-brain barrier. An association between QSM rim+ lesions and the therapeutic effect of cladribine could help select a subgroup of patients most likely to benefit from anti-inflammatory treatments. The measurement of serum biomarkers will enable an assessment of the activation of the peripheral immune system (cytokine, chemokines) and of the therapeutic effect of cladribine (NfL, GFAP). The positive results of the current project will allow the design of a phase 3 trial. A practical benefit of the proposed study is that patients with SPSM, who are currently not eligible for any treatment options, will have a choice to receive a potentially effective therapy, which costs substantially less compared to other therapies in MS.

Background: Multiple sclerosis (MS) is the most common chronic inflammatory, demyelinating disease of the central nervous system, with about 2.5 million patients worldwide, including 45 thousand in Poland. Most patients have relapsing-remitting MS (RRMS) at the start of the disease, in which neurological symptoms appear during relapses and may subside. There is a dozen of disease-modifying treatments for this form of the disease. Several years after the diagnosis of RRMS, the disease progresses into SPMS, in which disability worsens gradually independently of relapses. Patients with SPMS suffer from restricted mobility (need walking aids, wheelchair), cognitive impairment, (difficulties in workplace and in managing everyday life), depression, pain due to spasticity, chronic fatigue, lack of sphincter control, or sexual dysfunction. These patients need more medical help (office visits, rehabilitation, hospitalization), are more often unemployed, and have a lower quality of life than do patients with RRMS. Currently, three disease-modifying treatments are available for patients with SPMS in Europe: interferon beta-1b (low efficacy), mitoxantrone (serious adverse effects), and siponimod. However, these medications can be used only in patients with active disease, i.e., in those with still observed relapses or active brain lesions on magnetic resonance imaging. Therefore, about a half of patients with SPMS cannot receive any disease-modifying treatment. The current understanding of the pathogenesis of MS suggests that there are two types of neuroinflammation since disease onset. Type-1 neuroinflammation is characterized by an acute, focal infiltration of pathogenic lymphocytes and autoantibodies, which is associated with blood-brain barrier disruption. This type of neuroinflammation may be responsible for relapses and contrast-enhancing lesions. Type-2 neuroinflammation is a chronic, smoldering process that takes place behind a closed blood-brain barrier, and it is characterized by slowly expanding lesions and follicle-like lymph structures in the meninges, and diffuse inflammatory changes in white matter and cortex. Other characteristics of type-2 neuroinflammation include microglial and astroglial activation, delayed maturation of oligodendrocytes, and inhibition of remyelination. These processes cause disease progression independently of relapses. Both types of neuroinflammation occur simultaneously since disease onset, but type-2 neuroinflammation is thought to predominate in the secondary progressive phase. Standard neuroimaging methods cannot pinpoint lesions that are specific for type 2 neuroinflammation, but longitudinal brain atrophy and enlargement of lesions can indirectly measure its magnitude. Quantitative susceptibility mapping (QSM), a new imaging technique, can indicate chronic inflammatory lesions that are surrounded by active microglia at the lesion border. Microglia because of iron load form a hypointense rim, and might be thus shown by QSM technique (rim+ lesions). However, QSM is not currently used in clinical practice it is now recommended for use in clinical trials.

The currently available disease modifying-treatments for SPMS act solely or mainly on type-1 neuroinflammation, and because of that they are approved for patients with relapses or active lesions only. Cladribine is approved for the treatment of RRMS. Cladribine substantially decreases the number of contrast-enhancing lesions and relapse frequency in patients with RRMS (an effect on type-1 neuroinflammation). Cladribine may also act on type-2 neuroinflammation i.e. on the autoreactive lymphocytes resident in the central nervous system, including tertiary lymphoid structures, because cladribine penetrates into the central nervous system through an intact blood-brain barrier. The effect on type-2 neuroinflammation is supported by the observation that oligoclonal bands disappear in patients with RRMS and SPMS after cladribine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of relapse-onset, secondary progressive multiple sclerosis based on the 2017 McDonald criteria
* Progression of disability over 24 months defined as an increase in the EDSS score of 1 or more for patients with EDSS ≤ 5.5 or of 0.5 or more for patients with EDSS > 5.5
* Lack of relapses over last 12 months
* EDSS of 3.5 - 7.5 inclusive
* Age of 30 - 65 years inclusive
* Duration of MS of 10 years or longer
* Pre-menopausal women must refrain from heterosexual intercourse or use a contraception method with a failure rate of < 1% from enrolment up to 6 months after the last dose of the investigational medicinal product
* Men must refrain from heterosexual intercourse from enrolment up to 6 months after the last dose of the investigational medicinal product or use a barrier method of contraception, with their female partners using a contraception method with a failure rate of <1%
* Able to fulfill all protocol requirements as judged by the investigator

Exclusion Criteria:

* Lack of written informed consent
* Previous cladribine treatment
* Hypersensitivity to the investigational medicinal product
* Eligible and willing to use interferon beta, siponimod, or mitoxantrone
* Unable to undergo magnetic resonance imaging
* Pregnancy or breastfeeding
* Does not agree to use contraception methods defined above
* Diseases of the nervous system, such as tumors, stroke, traumatic injury, encephalomyelitis, B12 deficiency, or demyelinating diseases other than multiple sclerosis
* Major comorbidities, such as cancer, liver failure, kidney failure, heart failure (NYHA II-III), or any other disease that may jeopardize patient safety or make it impossible for the patient to fulfill protocol requirements
* Relapse within last 12 months
* Chronic treatment with corticosteroids or immunosuppressants (eg, azathioprine, methotrexate, cyclosporine) within last 6 months
* Disease-modifying treatments for multiple sclerosis (no washout is required for interferons beta, glatiramer acetate, and dimethyl fumarate; washout of > 6 months for teriflunomide, fingolimod, and natalizumab [an accelerate elimination procedure may be used for teriflunomide instead]; washout of > 12 months for ocrelizumab, mitoxantrone, and alemtuzumab)
* Relapsing-remitting multiple sclerosis
* Primary progressive multiple sclerosis
* Hepatitis B or hepatitis C, including detectable HbsA, anti-HBc, or anti-HCV antibodies in serum
* HIV infection, including a positive screening test (anti-HIV 1/2, protein 24)
* Active or latent tuberculosis, including a positive result of the QuantiFERON TB Gold test during screening or within 3 months (an inconclusive test must be repeated; two inconclusive tests are taken as a positive result)
* Other infection that may be worsened by treatment with cladribine
* Lymphopenia (< 1000/μl), neutrocytopenia (< 1500/μl), or thrombocytopenia
* Alanine aminotransferase or aspartate aminotransferase > 2 x ULN (can be repeated when 1.5-3x ULN); Total bilirubin > 1.5 x ULN (can be repeated when 1.5-3 x ULN); Hemoglobin > 9.5 g/dL (can be repeated when 9-9.4 g/dL)
* Lack of vaccination against COVID-19 - the time from the last dose of a full vaccination regimen is shorter than 6 weeks
* Any vaccination within last 6 weeks
* Lack of cancer screening or suspicion of cancer or necessity to carry out additional studies after the following examinations done at screening: chest X-ray in all participants; mammography or breast ultrasound in women; cervical smear in women; prostate-specific antigen in men
* Patient does not have detectable antibodies against Varicella zoster virus in serum or a proof of two-dose vaccination against this virus (last dose at least 6 months before enrolment)
* Use of oral or parenteral anticoagulants or antiplatelets other than acetylsalicylic acid

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Percent brain volume | 26 week following baseline
  brain volume to total intracranial volume
Percent brain volume | 122 week following baseline
  brain volume to total intracranial volume

SECONDARY OUTCOMES:
24 weeks confirmed composite progression of disability | 96 week
  Time to 24-week confirmed composite progression of disability defined as the occurrence of any of the following events: (1) an increase in the EDSS score of 1 or greater in patients with baseline EDSS ≤ 5.5 or of 0.5 or greater in those with baseline EDSS > 5.5; (2) an increase of 20% or more in Timed 25-Foot Walk; (3) an increase of 20% or more in the 9-Hole Peg Test.
Symbol-Digit Modality Test | 26 week
  Cognitive performance assessed with Symbol-Digit Modality Test
Symbol-Digit Modality Test | 96 week
  Cognitive performance assessed with Symbol-Digit Modality Test
California Verbal Learning Test | 26 week
  Cognitive performance assessed with California Verbal Learning Test [Polish version 2010]
California Verbal Learning Test | 122 week
  Cognitive performance assessed with California Verbal Learning Test [Polish version 2010]
Multiple Sclerosis Quality of Life Questionnaire 54 [MSQOL-54] | 26 week
  The MSQOL-54 is a structured, self-report questionnaire filled by the patient.The 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The summary scores are the physical health composite summary and the mental health composite summary, each may achieve final score from 0 to 100 points.
Multiple Sclerosis Quality of Life Questionnaire 54 [MSQOL-54] | 122 week
  The MSQOL-54 is a structured, self-report questionnaire filled by the patient.The 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The summary scores are the physical health composite summary and the mental health composite summary, each may achieve final score from 0 to 100 points.
Assessment of disease activity in MRI | 96 week
  Number of Gd+ lesions Number of new/enlarging T2 lesions
Assesment of chronic inflammation in MRI | 96 week
  Number of QSM rim+ lesions
Volume change of cervical spine | 96 week
  Volume of cervical spinal cord in T1
Laboratory measures -neurofilament light chain serum level | 0 to 122 week
  Concentration of neurofilament light chain in serum
Laboratory measures | 0 to 122 week
  Concentration of GFAP in serum
Laboratory measures - pro-inflammatory cytokines | 0 to 122 week
  Concentration of cytokines in serum
Oligoclonal bands (OCB) | 0 to 122 week
  Presence of oligoclonal bands in cerebrospinal fluid (selected patients who will sign an additional consent)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Kurkowska-Jastrzebska, MD, PhD, Principal Investigator — Institute for Psychiatry and Neurology
Locations (1):
- Institute of Psychiatry and Neurology, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lassmann H. Pathogenic Mechanisms Associated With Different Clinical Courses of Multiple Sclerosis. Front Immunol. 2019 Jan 10;9:3116. doi: 10.3389/fimmu.2018.03116. eCollection 2018. PMID 30687321
- [Background] Jamroz-Wisniewska A, Beltowski J, Wojcicka G, Bartosik-Psujek H, Rejdak K. Cladribine Treatment Improved Homocysteine Metabolism and Increased Total Serum Antioxidant Activity in Secondary Progressive Multiple Sclerosis Patients. Oxid Med Cell Longev. 2020 Mar 14;2020:1654754. doi: 10.1155/2020/1654754. eCollection 2020. PMID 32256946
- [Background] Fox RJ, Chataway J. Advancing trial design in progressive multiple sclerosis. Mult Scler. 2017 Oct;23(12):1573-1578. doi: 10.1177/1352458517729768. PMID 29041871
- [Background] Meinl E, Krumbholz M, Derfuss T, Junker A, Hohlfeld R. Compartmentalization of inflammation in the CNS: a major mechanism driving progressive multiple sclerosis. J Neurol Sci. 2008 Nov 15;274(1-2):42-4. doi: 10.1016/j.jns.2008.06.032. Epub 2008 Aug 19. PMID 18715571
- [Background] Montalban X, Belachew S, Wolinsky JS. Ocrelizumab in Primary Progressive and Relapsing Multiple Sclerosis. N Engl J Med. 2017 Apr 27;376(17):1694. doi: 10.1056/NEJMc1702076. No abstract available. PMID 28445663
- [Background] Comi G, Cook S, Giovannoni G, Rieckmann P, Sorensen PS, Vermersch P, Galazka A, Nolting A, Hicking C, Dangond F. Effect of cladribine tablets on lymphocyte reduction and repopulation dynamics in patients with relapsing multiple sclerosis. Mult Scler Relat Disord. 2019 Apr;29:168-174. doi: 10.1016/j.msard.2019.01.038. Epub 2019 Jan 24. PMID 30885375
- [Background] Liliemark J. The clinical pharmacokinetics of cladribine. Clin Pharmacokinet. 1997 Feb;32(2):120-31. doi: 10.2165/00003088-199732020-00003. PMID 9068927
- [Background] Sipe JC, Romine JS, Koziol JA, McMillan R, Zyroff J, Beutler E. Cladribine in treatment of chronic progressive multiple sclerosis. Lancet. 1994 Jul 2;344(8914):9-13. doi: 10.1016/s0140-6736(94)91046-4. PMID 7912347
- [Background] Rejdak K, Stelmasiak Z, Grieb P. Cladribine induces long lasting oligoclonal bands disappearance in relapsing multiple sclerosis patients: 10-year observational study. Mult Scler Relat Disord. 2019 Jan;27:117-120. doi: 10.1016/j.msard.2018.10.006. Epub 2018 Oct 10. PMID 30368223
- [Background] Jorgensen LO, Hyrlov KH, Elkjaer ML, Weber AB, Pedersen AE, Svenningsen AF, Illes Z. Cladribine modifies functional properties of microglia. Clin Exp Immunol. 2020 Sep;201(3):328-340. doi: 10.1111/cei.13473. Epub 2020 Jul 6. PMID 32492189
- [Background] Montalban X, Gold R, Thompson AJ, Otero-Romero S, Amato MP, Chandraratna D, Clanet M, Comi G, Derfuss T, Fazekas F, Hartung HP, Havrdova E, Hemmer B, Kappos L, Liblau R, Lubetzki C, Marcus E, Miller DH, Olsson T, Pilling S, Selmaj K, Siva A, Sorensen PS, Sormani MP, Thalheim C, Wiendl H, Zipp F. ECTRIMS/EAN Guideline on the pharmacological treatment of people with multiple sclerosis. Mult Scler. 2018 Feb;24(2):96-120. doi: 10.1177/1352458517751049. Epub 2018 Jan 20. PMID 29353550
- [Background] Frischer JM, Weigand SD, Guo Y, Kale N, Parisi JE, Pirko I, Mandrekar J, Bramow S, Metz I, Bruck W, Lassmann H, Lucchinetti CF. Clinical and pathological insights into the dynamic nature of the white matter multiple sclerosis plaque. Ann Neurol. 2015 Nov;78(5):710-21. doi: 10.1002/ana.24497. Epub 2015 Aug 24. PMID 26239536
- [Background] Hametner S, Wimmer I, Haider L, Pfeifenbring S, Bruck W, Lassmann H. Iron and neurodegeneration in the multiple sclerosis brain. Ann Neurol. 2013 Dec;74(6):848-61. doi: 10.1002/ana.23974. Epub 2013 Oct 7. PMID 23868451
- [Background] Dal-Bianco A, Grabner G, Kronnerwetter C, Weber M, Hoftberger R, Berger T, Auff E, Leutmezer F, Trattnig S, Lassmann H, Bagnato F, Hametner S. Slow expansion of multiple sclerosis iron rim lesions: pathology and 7 T magnetic resonance imaging. Acta Neuropathol. 2017 Jan;133(1):25-42. doi: 10.1007/s00401-016-1636-z. Epub 2016 Oct 27. PMID 27796537
- [Background] Absinta M, Sati P, Masuzzo F, Nair G, Sethi V, Kolb H, Ohayon J, Wu T, Cortese ICM, Reich DS. Association of Chronic Active Multiple Sclerosis Lesions With Disability In Vivo. JAMA Neurol. 2019 Dec 1;76(12):1474-1483. doi: 10.1001/jamaneurol.2019.2399. PMID 31403674
- [Background] Kaunzner UW, Kang Y, Zhang S, Morris E, Yao Y, Pandya S, Hurtado Rua SM, Park C, Gillen KM, Nguyen TD, Wang Y, Pitt D, Gauthier SA. Quantitative susceptibility mapping identifies inflammation in a subset of chronic multiple sclerosis lesions. Brain. 2019 Jan 1;142(1):133-145. doi: 10.1093/brain/awy296. PMID 30561514
- [Background] Elliott C, Wolinsky JS, Hauser SL, Kappos L, Barkhof F, Bernasconi C, Wei W, Belachew S, Arnold DL. Slowly expanding/evolving lesions as a magnetic resonance imaging marker of chronic active multiple sclerosis lesions. Mult Scler. 2019 Dec;25(14):1915-1925. doi: 10.1177/1352458518814117. Epub 2018 Dec 19. PMID 30566027
- [Background] Wang CT, Barnett M, Barnett Y. Imaging the multiple sclerosis lesion: insights into pathogenesis, progression and repair. Curr Opin Neurol. 2019 Jun;32(3):338-345. doi: 10.1097/WCO.0000000000000698. PMID 30950846